CLINICAL TRIAL: NCT07119996
Title: A Phase Ib Study Evaluating the Safety and Efficacy of Vitamin B3 Combined With Neoadjuvant Tislelizumab Plus Gemcitabine/Cisplatin in Antibiotic-Exposed Patients With cT2-T4aN0M0 Urothelial Carcinoma of the Bladder
Brief Title: Clinical Trial on the Protective Role of Vitamin B3 in Enhancing Immunotherapy for Bladder Cancer Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-20241202
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer
Keywords: Antibiotics; Nicotinamide nucleotides; Immunotherapy; Bladder Cancer
MeSH Terms: conditions — Neoplasms; Urinary Bladder Neoplasms | interventions — tislelizumab; Cisplatin; Gemcitabine; Niacinamide; Niacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin B3 supplement (Experimental): Arm Description: During each 21 days study cycle(up to 6 cycles), all participants will receive: a) Tislelizumab: Taken 1x time at d1 each cycle or until it is determined participant must stop the drug. b) Gemcitabine: d1, d8 each cycle or until it is determined participant must stop the drug. c) Cisplatin: d2 each cycle or until it is determined participant must stop the drug. Tislelizumab maintenance therapy:after chemoimmunotherapy, q3W until it is determined participant must stop the drug, or 2 years of treatment is completed. d) Oral Vitamin B3 supplementation (2 predefined dose) intake
  Interventions: Drug: Tislelizumab, Cisplatin, Gemcitabine and Vitamin B3

INTERVENTIONS:
Drug: Tislelizumab, Cisplatin, Gemcitabine and Vitamin B3 — 1. Tislelizumab: 200mg, 1x time at d1 each cycle
  2. Gemcitabine: 1000mg/ m2, in d1, d8 each cycle
  3. Cisplatin: 70 mg/m2, in d2 each cycle Tislelizumab maintenance therapy: after chemoimmunotherapy, 200mg, q3W.
  4. Vitamin B3 tablet(also known as nicotinic acid tablet) supplementation daily(300mg QD or 500mg QD) after antibiotic treatment.
  Other Names: Nicotinic Acid Tablets; Tislelizumab; Cisplatin; Gemcitabine

SUMMARY:
When bladder cancer patients are treated to mobilize their own immune system to fight the tumor, drugs that kill the bacteria can impair the effectiveness of the treatment. The purpose of this study is to find out if the common dietary supplement Vitamin B3 could allow drugs that kill bacteria to not negatively affect treatments that mobilize the immune system to fight tumors.

ELIGIBILITY:
Inclusion Criteria

1. The patient voluntarily agrees to participate, is able to provide written informed consent, and is willing and able to comply with the protocol and schedule of assessments.
2. Aged ≥18 years on the date of signing the informed-consent form (ICF).
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Appendix 1).
4. Residual tumour after TURBT and histologically confirmed urothelial carcinoma of the bladder staged cT2-T4a N0 M0 by AJCC 8th edition imaging; for mixed-histology tumours, the urothelial component must be predominant (≥50 %).
5. An infection occurring from 30 days to 1 day before the first dose of immuno-chemotherapy that, in the judgement of the attending physician, required oral or intravenous bactericidal antibiotics and met any of the following diagnostic criteria:

   1. Clinical features (e.g. ≥38.3 °C or sustained ≥38 °C for ≥1 h with chills, local pain, dysuria, etc.) plus laboratory evidence (WBC > 10 × 10⁹/L or < 4 × 10⁹/L, neutrophilia / neutropenia, markedly elevated CRP) consistent with bacterial infection;
   2. Abnormal urinalysis suggestive of urinary-tract infection (e.g. WBC > 10/HPF, bacteria seen on high-power field, nitrite positive) with pathogen confirmed by urine culture;
   3. Infection confirmed by imaging or other microbiological tests (e.g. blood culture, nasopharyngeal swab, sputum culture).

   Permitted bactericidal antibiotics (oral or IV) include but are not limited to:
   1. β-lactams (penicillins, cephalosporins, carbapenems);
   2. Glycopeptides (vancomycin, teicoplanin);
   3. Quinolones (levofloxacin, ciprofloxacin);
   4. Aminoglycosides (gentamicin, streptomycin).
6. Adequate organ function, documented within ≤14 days before enrolment:

   a. No growth-factor support ≤14 days before sampling and: i. Absolute neutrophil count ≥1.5 × 10⁹/L; ii. Platelets ≥90 × 10⁹/L; iii. Haemoglobin ≥90 g/L; b. INR or aPTT ≤1.5 × ULN; c. Total bilirubin ≤1.5 × ULN (≤3 × ULN for Gilbert's syndrome or isolated indirect hyper-bilirubinaemia of extra-hepatic origin); d. AST, ALT and alkaline phosphatase ≤2.5 × ULN; e. Pulmonary function adequate to tolerate major abdominal surgery.
7. Considered cisplatin-eligible by the investigator. Patients deemed cisplatin-ineligible must meet ≥1 of: ECOG > 1 or Karnofsky 60-70 %; creatinine clearance < 60 mL/min; NCI-CTCAE v5.0 grade ≥2 hearing loss; NCI-CTCAE v5.0 grade ≥2 peripheral neuropathy; New York Heart Association class III or IV heart failure.
8. Women of child-bearing potential agree to use highly effective contraception during the study and for ≥120 days after the last dose of tislelizumab or chemotherapy (whichever is later) and have a negative urine or serum pregnancy test ≤7 days before enrolment. Non-sterilised men likewise agree to use highly effective contraception for the same period (Appendix 5).

Exclusion Criteria

Patients meeting any of the following are ineligible:

1. Previous therapy directed against PD-1, PD-L1, PD-L2, CTLA-4 or any other antibody or drug targeting T-cell co-stimulation or checkpoint pathways.
2. Systemic anticancer therapy or systemic immunomodulator (e.g. interferon, interleukin-2, TNF) within 28 days before enrolment.
3. Prior radiotherapy to the bladder.
4. Prior antitumour drug therapy, except:

   1. ≥12 months since the last dose of systemic chemotherapy before study neoadjuvant therapy;
   2. Intravesical chemotherapy or immunotherapy completed ≥1 week before study treatment.
5. Major surgery or significant trauma within 28 days before enrolment (vascular-access placement and TURBT are not major surgery).
6. Live vaccine within 28 days before enrolment (inactivated seasonal influenza vaccine is permitted; intranasal influenza vaccine is live and prohibited).
7. Active autoimmune disease requiring systemic therapy that, in the investigator's opinion, would interfere with study treatment.
8. Long-term high-dose corticosteroids or other immunosuppressants that, in the investigator's opinion, would interfere with study treatment.
9. Clinically significant abnormalities that could affect treatment, including electrolyte disturbance (K, Na, Ca), hypoalbuminaemia, interstitial lung disease, non-infectious pneumonitis, or other uncontrolled systemic diseases (e.g. diabetes, hypertension, cardiovascular disease such as severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, or clinically significant ventricular arrhythmia within 6 months).
10. Untreated chronic HBV infection with HBV-DNA ≥500 IU/mL (2,500 copies/mL) or HBsAg carrier status. Patients with inactive HBsAg carriage or stable active HBV on antiviral therapy with HBV-DNA < 500 IU/mL may enrol. HBV-DNA testing is required only for anti-HBc-positive patients.
11. Active HCV infection. Patients who are anti-HCV-negative, or anti-HCV-positive but HCV-RNA-negative, may enrol. Anti-HCV-positive patients must have HCV-RNA testing.
12. History of immunodeficiency (including HIV positivity or other acquired/congenital immunodeficiencies), or prior allogeneic stem-cell or solid-organ transplantation (Appendix 3).
13. Known hypersensitivity to other monoclonal antibodies.
14. Known hypersensitivity to any study drug or excipient.
15. Unresolved toxicities from prior therapy that have not returned to baseline or stabilised, unless considered by the investigator not to pose a safety risk (e.g. alopecia, neuropathy, certain laboratory abnormalities).
16. Any condition (medical or substance abuse) that could impede study-drug administration, confound interpretation of results, or place the patient at high risk of complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: The DLT dose of the Vitamin B3 | 28 days after the first dose (D1-D28)
  Participants with dose-limiting toxicity (DLT) asassessed by NCl CTC 5.0 and the administered drug dose.

SECONDARY OUTCOMES:
Percentage of Participants With Pathological Downstaging(pDS) | 24 Months
  The pathological downstaging rate is defined as the evaluation of whether the staging is degraded to ≤ T2 based on the post-surgery pathological findings. The rates of cT2N0 → pT0N0, cT3-4aN0 → pT0N0, cT2N0 → ≤ pT1N0, cT3-4aN0 → ≤ pT1N0 will be calculated, and the 2 sided Clopper-Pearson 95% confidence interval (CI) of pathological downstaging rate will be calculated to assess the precision of the estimated pathological downstaging rate.
Safety and AE | 24 months
  Number of unique patients who had a treatment-related (possible, probable, or definite) adverse event using the Medical Dictionary for Regulatory Activities (MedDRA) terms and graded per NCI-CTCAE v5.0. Number and Grade of patients who had a surgery-related adverse event (surgery-related AE) will be measured according to the Clavien-Dindo classification.
Percentage of Participants With Pathological Complete Response(pCR) | 24 months
  Pathological evaluation of the resected tumor tissue and regional lymph nodes showed no residual tumor cells, complete disappearance of the tumor lesions, and no evidence of new lesions.

OTHER OUTCOMES:
Biomarker Endpoint Analyses | 24 months
  To explore biomarkers in urine, blood, and tumor tissues (collected from TURBT) atbaseline and tissue samples collected from radical cystectomy. Biomarkers include PD-L1, Mki67 expression in tumor tissues, immune cells profling and gene expression and tumor mutation profiling.

CONTACTS AND LOCATIONS:
Overall Officials: Tianxin Lin, Ph.D, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: Undecided